CLINICAL TRIAL: NCT01675856
Title: Urgent vs. Early Endoscopy in High Risk Patients With UGIB
Brief Title: Urgent vs. Early Endoscopy in High Risk Patients With Upper Gastrointestinal Bleeding (UGIB)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, James Yun-wong Lau, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AUGIB
Record Dates: First submitted 2012-08-27; First posted 2012-08-30 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Bleeding Peptic Ulcer; Active Bleeding; Gastrointestinal Bleeding
Keywords: Glasgow-Blatchford score; Gastrointestinal bleeding
MeSH Terms: conditions — Peptic Ulcer Hemorrhage; Gastrointestinal Hemorrhage

STUDY DESIGN:
Intervention Model Description: Patients are randomized in a 1:1 ratio. The patient is randomized to receive;
  1. Urgent endoscopy (defined by endoscopy within 6 hours from first consultation by GI specialists at PWH) or
  2. Early endoscopy (defined by endoscopy next morning and within 24 hours from first consultation by GI specialists at PWH)
Oversight: Data Monitoring Committee: No

ARMS (2):
- Urgent endoscopy (Active Comparator): Oesophagogastroduodenoscopy done within 6hours of first GI specialists consultation
  Interventions: Other: Urgent endoscopy
- Early endoscopy (Placebo Comparator): Oesophagogastroduodenoscopy done within 24hours of first GI specialists consultation
  Interventions: Other: Early endoscopy

INTERVENTIONS:
Other: Urgent endoscopy — Defined by oesophagogastroduodenoscopy within 6 hours of first presentation of Prince of Wales Hospital
  Arms: Urgent endoscopy
Other: Early endoscopy — Defined by oesophagogastroduodenoscopy within 24 hours of first presentation of Prince of Wales Hospital
  Arms: Early endoscopy

SUMMARY:
Acute upper gastrointestinal bleeding (UGIB) is one of the commonest medical emergencies. The condition accounts for 150 per 100,000 populations. A National United Kingdom reported a crude overall mortality rate of 10%. While bleeding stops spontaneously in majority of patients at their presentation, there remains a subgroup of patients who continue to bleed or develop recurrent bleeding. In these patients, the mortality increases manifolds. If these high-risk patients can be identified, early interventions may improve their outcomes.

Several prognostic indices are in use for the purpose of patient stratification. They include the Rockall, Glasgow-Blatchford (GBS) and the Baylor scores. The Rockall score is a composite score which incorporates clinical parameters as well as findings during endoscopy which was derived to predict mortality. The GBS is a pre-endoscopy or a clinical score for the prediction for the need of further intervention loosely defined as the need for transfusion, endoscopy or surgery. It has been shown to be accurate in identifying low risk patients for early discharge.

DETAILED DESCRIPTION:
The GBS, being a pre-endoscopy score with clinical parameters, is more suitable for patient triage leading to urgent endoscopy and a higher level of care. A GBS of 0 has been shown to identify patients with upper gastrointestinal bleeding who may be managed safely as outpatients. The proportion of patients requiring endoscopic therapy increases with a higher score. A cut-off score that identifies "high-risk" patients who may benefit from urgent intervention however has not been determined. Guidelines from Societies around the world recommend early endoscopy within 24 hours of presentation for acute upper gastrointestinal bleeding (AUGIB). The guidelines also state that a proportion of patients need emergency "out-of-hours" endoscopy, without defining the "high-risk" group. A recent international consensus on the management of NVUGIB recommended early endoscopy within 24 hours for Non-Variceal Upper Gastro Intestinal Bleeding (NVUGIB), and noted no additional benefit associated with urgent endoscopy (<12 hours) vs. early endoscopy (>12 hours) in unselected patients with NVUGIB. However, there are only limited data on the role of urgent endoscopy in the "selected" subgroup of patients with high-risk NVUGIB.

ELIGIBILITY:
Inclusion Criteria:

1. Overt signs of upper gastrointestinal bleeding (i.e., melena or hematemesis with or without hypotension)
2. GBS of ≥12
3. In-patients admitted for reasons other than AUGIB who develop bleeding are also considered for trial enrollment.
4. Patients in Hypotensive shock (SBP ≤90 mmHg or pulse ≥110 bpm) are initially resuscitated and then considered for trial entry if their condition can be stabilized.

Exclusion Criteria:

1. continued shock despite initial volume resuscitation (refractory shock) undergo urgent endoscopy
2. < 18 years of age
3. Unable to provide written informed consent
4. Pregnant or lactating women
5. Moribund patients from terminal illnesses. (active treatment not considered)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2012-07-28 (Actual); Primary Completion 2018-11-11 (Actual); Study Completion 2018-11-11 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 days
  Death from all causes 30 days from randomization

SECONDARY OUTCOMES:
Need for endoscopic therapy at index endoscopy | At the time of index endoscopy
  To measure if endoscopic therapy is needed at the index endoscopy
Need for transfusion | Within 30days of randomization
  To measure if transfusion of blood products is needed within 30days of randomization
Recurrent bleeding as defined | Within 30days of randomization
  To measure if any clinical or endoscopic recurrent bleeding is identified.
Duration of hospital stay of index bleeding | Within 30 days of randomization
  To measure the number of days of hospital stay upon randomization, only counted the hospitalization days of index bleeding.
ICU stay | Within 30days of randomization
  To measure if ICU admission is required at the index bleeding.
Need for further endoscopic treatment | Within 30days of randomization
  To measure if further endoscopic treatment if required at recurrent bleeding
Emergency surgery or interventional radiology to achieve hemostasis | Within 30days of randomization
  To measure if emergency surgery or interventional radiology is needed at index bleeding or recurrent bleeding to achieve hemostasis
Rates of recurrent bleeding | Within 30 days of randomization
  To measure recurrent bleeding in both study arms
Rate of adverse events | Within 30 days of randomization
  To measure the adverse events in either group, e.g. myocardial event, cerebrovascular event and acute renal failure.

CONTACTS AND LOCATIONS:
Overall Officials: James Y LAU, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Endoscopy Centre, Prince of Wales Hospital, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lau JYW, Yu Y, Tang RSY, Chan HCH, Yip HC, Chan SM, Luk SWY, Wong SH, Lau LHS, Lui RN, Chan TT, Mak JWY, Chan FKL, Sung JJY. Timing of Endoscopy for Acute Upper Gastrointestinal Bleeding. N Engl J Med. 2020 Apr 2;382(14):1299-1308. doi: 10.1056/NEJMoa1912484. PMID 32242355